CLINICAL TRIAL: NCT03243877
Title: Multi-Centric Screening of Breast Cancer Patients to Determine Efficiency and to Assess Sensitivity & Accuracy of Pandora CDx MammoAlertTM in Screening of Breast Cancer.
Brief Title: Performance of MammoAlert™, Point of Care System, for the Screening of Breast Cancer in Women 18 Years of Age or Older
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: POC Medical Systems, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: POC-BC-0217
Record Dates: First submitted 2017-07-25; First posted 2017-08-09 (Actual); Last update posted 2018-04-11 (Actual); Status verified 2018-04

CONDITIONS: Breast Cancer
Keywords: Screening; Mammography
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Breast Cancer Positive: A 5cc blood sample will be collected from subjects who were screened for breast cancer at the treating facility and results were positive.
  MammoAlert Screening Test will be performed on plasma obtained from the blood sample.
  Interventions: Other: MammoAlert Screening Test
- Breast Cancer Negative: A 5cc blood sample will be collected from subjects who were screened for breast cancer at the treating facility and results were negative.
  MammoAlert Screening Test will be performed on plasma obtained from the blood sample.
  Interventions: Other: MammoAlert Screening Test

INTERVENTIONS:
Other: MammoAlert Screening Test — Plasma obtained from blood samples will be analyzed with the MammoAlert Screening Test for the presence of known breast cancer bio-markers.

SUMMARY:
POC Medical Systems has developed a Point of Care system for the screening of breast cancer in the general population. Via a proprietary algorithm, the MammoAlert™ is expected to determine breast cancer's risk level for a subject by identifying the presence in plasma of known biomarkers. The present study aims to determine the Sensitivity and Specificity of the test in plasma samples of subjects of whom the status vis-à-vis breast cancer is known.

DETAILED DESCRIPTION:
2400 subjects will be screened for breast cancer in seven enrolling sites across the country to ensure diverse ethnicity.

"Positive" subjects should be confirmed breast cancer positive by Mammography and/or biopsy. Breast cancer positive samples will be compared to the control group of samples obtained from women attending clinics for non-cancerous related pathology.

Both Positive and Negative Predictive Values will be evaluated to determine accuracy and sensitivity of the screening test.

Subjects whose known cancer positive or negative status do not match the test report will be followed up as appropriate, on case by case basis to identify false positive and false negative results.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to give informed consent. Written informed consent by the patient/patient's legally acceptable representative (LAR) for donating blood sample
2. Documented absence of cancer (other than Breast Cancer)
3. Documented (Mammography and/or Biopsy) diagnosis of Breast Cancer (IDC/ILC/DCIS ), any stage
4. Blood sample taken before any treatment for Breast Cancer was administered to the subject.

Exclusion Criteria:

1. Other malignancy besides breast cancer in the 5 years prior to obtaining the sample.
2. Therapies for breast cancer that have been administered within 1 year of obtaining the sample
3. Any condition (including psychiatric), which in the Investigator's opinion, places the patient at undue risk by participating in the study.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Gender Based: Yes — Women only
Study Population: The present study targets women of at least 18 years old
Sampling Method: Probability Sample
Enrollment: 2458 (Actual)
Dates: Start 2017-06-17 (Actual); Primary Completion 2017-11-26 (Actual); Study Completion 2018-08-31 (Estimated)

PRIMARY OUTCOMES:
Screening performance (i.e., sensitivity and specificity) | Screening performance will be calculated at 4-months
  Screening performance: comprises the sensitivity and specificity of MammoAlert™. It represents the performance of the diagnostic test and is therefore independent of the prevalence of the disease in the studied sample of patients.

SECONDARY OUTCOMES:
Predictive values & likelihood ratios | Predictive values & likelihood ratios will be calculated at 4-months
  Positive predictive value: the probability that a subject has the disease given that the test result is positive will be estimated by: TP/(TP+FP).
  Negative predictive value: the probability that a subject does not have the disease given that the result of the test is negative will be estimated by TN/(TN+FN).
  Likelihood ratio (LR): the likelihood that a given test result would be expected in a patient with the target disorder compared to the likelihood that that same result would be expected in a patient without the target disorder.

OTHER OUTCOMES:
Accuracy of test | Accuracy of test will be calculated at 4-months
  The probability that the test result reflects the true disease state will be estimated as the proportion of cases for which the test result is correct: (TP+TN)/(TP+FP+TN+FN).
Reproducibility | Reproducibility will be calculated at 4-months
  The ability of MammoAlert™ to reveal the same result when repeatedly performed on the same sample, assessed repeatedly by the same reader

CONTACTS AND LOCATIONS:
Overall Officials: Raghu Ram Pillarisetti, MD, Principal Investigator — KIMS USHALAKSHMI Centre for Breast Diseases KIMS Hospitals
Locations (7):
- India (7):
  - KIMS USHALAKSHMI Centre for Breast Diseases KIMS Hospitals, Hyderabad, Andhra Pradesh
  - Indo American Cancer Hospital and Research Institute, Hyderabad, Andhra Pradesh
  - HCG MULTI Specialty Hospital HCG Cancer Center, Ahmedabad, Gujarat
  - Manipal Hospital, Bangalore, Karnataka
  - Amrita Institute of Medical Sciences and Research Centre, Kochi, Kerala
  - Tata Medical Center, Kolkata, West Bengal
  - Maulana Azad Medical College University of Delhi & Associated Lok Nayak Hospital, New Delhi

IPD SHARING:
Plan to Share IPD: No